CLINICAL TRIAL: NCT04843709
Title: An Open-Label, Multi-center, Phase I/II Dose Escalation and Expansion Study to Assess the Safety, Tolerability, Anti-Tumor Activity and Pharmacokinetics of MRG004A in Patients With Tissue Factor Positive Advanced or Metastatic Solid Tumors
Brief Title: A Study of MRG004A in Patients With Tissue Factor Positive Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG004A-001
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Advanced or Metastatic Solid Tumors
Keywords: MRG004A; Antibody drug conjugate (ADC); Tissue factor; Solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MRG004A (Experimental): All patients in Part A (dose escalation) and Part B (dose expansion) will be administrated MRG004A on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG004A

INTERVENTIONS:
Drug: MRG004A — Administrated intravenously

SUMMARY:
The objective of this study is to evaluate the safety, efficacy, pharmacokinetics, and immunogenicity of MRG004A in patients with Tissue Factor positive advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This study consists of two parts. Part A is a dose escalation study to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of MRG004A. Part B is a disease specific multi-cohort dose expansion study to further assess the efficacy and safety of MRG004A at confirmed RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Understands and provides written informed consent and willing to follow the requirements specified in protocol.
2. Age ≥18 years.
3. Life expectancy ≥6 months.
4. For Part B patients, documented Tissue Factor (TF) presence in tumor biopsy specimens obtained from archival or re-biopsy specimens by immunohistochemistry (IHC) protein expression.
5. Must have histologically or cytologically confirmed unresectable or metastatic cancer with documented disease progression during prior therapy, or relapse or progression following approved standard therapy for their tumor types- Part A and Part B.
6. Part B: Patients who have documented progression during or relapse following standard therapy, no further treatment options that are known to improve survival, and participation in a clinical trial is a reasonable therapeutic option.
7. Patients must have measurable disease per RECIST v1.1.
8. ECOG performance status of 0 or 1.
9. Acceptable bone marrow, hepatic, cardiac, renal, and coagulation function.
10. A negative serum pregnancy test if female and aged between 18-55 years old.
11. Patients, both females and males, of reproductive potential must agree to use adequate contraception during and for 180 days after the last infusion of MRG004A.

Exclusion Criteria:

1. Archival or biopsy tumor shows TF IHC membrane or cytosolic score of zero, no TF-positive expression or no TF-positive staining in Part B patients.
2. Toxicities (except alopecia & fatigue) due to prior antitumor therapy are greater than CTCAE v5.0 Grade 1.
3. Toxicities due to prior radiotherapy that have not resolved to Grade ≤ 1 CTCAE v5.0 at least 21 days prior to the first treatment.
4. Untreated, unstable or uncontrolled central nervous system (CNS) metastases.
5. Any other type of anti-cancer therapy within 21 days of the first dose of study treatment. Use of any other type of anti-cancer treatment is prohibited throughout the study.
6. Patients with increased bleeding risk.
7. Presence of severe cardiac dysfunction.
8. Pulmonary embolism or deep vein thrombosis within 3 months prior to the first dose of study drug.
9. Concurrent malignancy within 5 years prior to entry.
10. Uncontrolled or poorly controlled hypertension.
11. History of ventricular tachycardia, or torsade des pointes.
12. History of moderate to severe dyspnea at rest.
13. Major surgery within 4 weeks of the first dose of study treatment and not fully recovered. Minor surgery within 2 weeks prior to study treatment.
14. Known allergic reactions to any component or excipient of MRG004A or known allergic reactions to other prior anti-TF (including investigational) or other monoclonal antibody ≥ Grade 3.
15. Patients who have any known liver disease, including chronic hepatitis B, hepatitis C, autoimmune hepatic disorders, primary biliary cirrhosis or sclerosing cholangitis; Patients who have concurrent, serious, uncontrolled infections or known infection with HIV, or have a diagnosed acquired immunodeficiency syndrome (AIDS); or an uncontrolled autoimmune disease, or have undergone organ transplant.
16. Active uncontrolled bacterial, viral, fungal, rickettsial, or parasitic infection.
17. Use of systemic corticosteroids within 4 weeks prior to the first dose of treatment.
18. Use of strong CYP3A4 inhibitors or inducers with MRG004A.
19. Other excluded medications or treatment: therapeutic anti-coagulative, or long-term anti-platelet treatment; multivitamins, calcium, vitamin D, and prophylactic anti-RANKL (denosumab) and zoledronic acid therapies for bone metastases are allowed.
20. Any patient with a positive pregnancy or is breast-feeding.
21. Any severe and/or uncontrolled systemic disease that at the discretion of investigator and sponsor makes it undesirable for the patient to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | DLT will be evaluated during the first treatment cycle (Day 1-21)
  The highest dose confirmed wherein less than 2 out of 6, or < 33% of evaluable patients in a treatment cohort experiences dose-limiting toxicity (DLT).
Recommended Phase II Dose (RP2D) | Baseline to study completion (up to 24 months)
  The dose level of MRG004A recommended for further clinical studies based on assessment of the safety, efficacy and PK data from Part A of this study.
Objective Response Rate (ORR) | Baseline to study completion (up to 24 months)
  The proportion of patients who achieve complete response (CR) or partial response (PR) as assessed by the Independent Central Review (ICR).
Adverse Events (AEs) | From signing informed consent until 45 days after the last dose of MRG004A
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.

SECONDARY OUTCOMES:
Duration of Response (DoR) | Baseline to study completion (up to 24 months)
  The time interval between the date of the earliest qualifying response and the date of disease progression or death for any cause, whichever occurs earlier.
Disease Control Rate (DCR) | Baseline to study completion (up to 24 months)
  The proportion of patients who achieve CR, PR, or stable disease (SD) ≥ 6 weeks based on RECIST v1.1.
Progression Free Survival (PFS) | Baseline to study completion (up to 24 months)
  The time from the date of first study dose to disease progression or death whichever occurs first.
Overall Survive (OS) | Baseline to study completion (up to 24 months)
  The time from start of study treatment to date of death as a result of any cause.
Pharmacokinetics (PK) Parameter of MRG004A: Cmax | Baseline to 30 days after the last dose of study treatment
  Maximum observed plasma concentration.
Pharmacokinetics (PK) Parameter of MRG004A: Tmax | Baseline to 30 days after the last dose of study treatment
  Time to reach the maximum plasma concentration.
Pharmacokinetics (PK) Parameter of MRG004A: AUClast | Baseline to 30 days after the last dose of study treatment
  Area under the plasma concentration-time curve from time 0 to the time of last quantifiable concentration.
Incidence of anti-drug antibody (ADA) | Baseline to 30 days after the last dose of study treatment
  The proportion of patients with positive ADA immunogenicity results.

CONTACTS AND LOCATIONS:
Overall Officials: Nashat Y Gabrail, MD, Principal Investigator — Gabrail Cancer Center Research
Locations (9):
- United States (6):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Memorial Sloan Kettering 60th Street Outpatient Center, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Virginia Cancer Specialists, Fairfax, Virginia
- China (3):
  - Hunan Cancer Hospital, Changsha, Hunan
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No